CLINICAL TRIAL: NCT03027544
Title: Tomotherapy for Refractory Brain Metastases: a Single Arm, Single Center Phase II Trial
Brief Title: Tomotherapy for Refractory Brain Metastases
Acronym: TRBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Dr, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2014 YZ-14
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Brain Metastases
Keywords: multiple brain metastases; large brain metastases; meningeal metastases; tomotherapy
MeSH Terms: conditions — Brain Neoplasms; Meningeal Carcinomatosis | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): Group A: multiple brain metastases: no less than 3 lesions in the brain Group B: Large Brain Metastases: the volume of lesion is no smaller than 6cc or the maximum diameter of the lesion is no shorter than 3cm Group C:Meningeal Metastases.
  Intervention：tomotherapy
  Interventions: Radiation: tomotherapy

INTERVENTIONS:
Radiation: tomotherapy — Tomotherapy: The regular fraction modes were as follows: a. lesions≥3 cm:52Gy/4Gy/13f or 52.5Gy/3.5Gy/15f; b. lesions<2cm:36Gy/12Gy/3f or 24Gy/24Gy/1f; for lesions located in function areas, it would be adjusted to 40Gy/8Gy/5f; c. lesions 2-3cm: 40-48Gy/8-10Gy/6-4f; d. lesions located in brainstem:50-60Gy/2.5-3Gy/20f; 3. multiple lesions with large lesion: whole brain radiation (WBRT) with 40Gy/2Gy/20f and concurrent boost of 60Gy/3Gy/20f of the lesions.
  TMZ is used if necessary: concomitant TMZ: 75mg/m2 adjuvant TMZ: 150mg/ m2*5d, q28d, up to 6cycles.

SUMMARY:
This clinical trial was designed to investigate the efficiency and toxicity of tomotherapy for refractory brain metastases.

DETAILED DESCRIPTION:
This is a single-arm, single center, phase II trial to investigate the feasibility and toxicity of tomotherapy for refractory brain metastases, which are defined as A: multiple brain metastases(≥3 lesions); B: large brain metastases(with one lesion's volume is no smaller than 6cc or the longest diameter is no shorter than 3cm); C: meningeal metastases.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of primary tumor and conformed brain metastases by enhanced MRI or CT; the lesion number is no less than 3; or the tumor volume is no smaller than 6cc; or tumor diameter is no shorter than 3cm; or uncontrolled brain tumor after whole brain radiotherapy(WBRT); or the tumor is adjacent to essential structures of the brain, such as brain stem, optic chiasma, optic tract, etc; KPS ≥60,or KPS ≥40 and the limitation of motion is simply caused by brain tumor that is adjacent to the motor function areas; Age: 18-75 years old;

Adequate end-organ function:

WBC≥4.0x109/L Neu ≥ 1.5x109/L Hemoglobin ≥ 110 g/L Platelets ≥100 x109/L Total bilirubin ≤ 1.5x ULN AST and ALT ≤ 1.5x ULN BUN and Cr: within the normal range.

Exclusion Criteria:

* • Other clinically significant diseases (e.g.myocardial infarction within the past 6 months, severe arrhythmia).

  * Unable or unwilling to comply with the study protocol.
  * The expected survival time is less than 3 months.
  * Patients who are anticipated in other clinical trials of brain metastases.
  * Patients who has been treated with SRT in other hospitals
  * Pregnant patients or female patients whose HCG is positive
  * Unsuitable to participate in study, that in the opinion of the treating physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2-3 months after radiation
  Using RTOG9508 criteria, Tumor control is defined as CR+PR+SD

SECONDARY OUTCOMES:
Overall survival rate | up to 3 years
progress free survival rate | up to 1 year
local control rate | up to 1 year
intracranial progress free survival rate | up to 1 year
adverse event | from the day of radiation, up to 6 months
cause of death | from the day of radiation to death date, up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Xiao, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
the baseline characteristics and treatment plan can be shared with other researchers when the research paper has been published. The IPD will be sent by email if applied.